CLINICAL TRIAL: NCT00663884
Title: A Prospective, Randomized and Multi-center Clinical Study to Evaluate Efficacy and Safety of Combination Therapy of Mitiglinide or Voglibose With Long-acting Insulin in Type 2 Diabetic Patients
Brief Title: Glufast On Insulin Glargine Trial in Type 2 DM
Acronym: GLORIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CWP-KAD-402
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, Type 2; mitiglinide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — mitiglinide; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M (Experimental): Mitiglinide
  Interventions: Drug: Mitiglinide
- V (Active Comparator): Voglibose
  Interventions: Drug: Voglibose

INTERVENTIONS:
Drug: Mitiglinide — mitiglinide 10mg three times a day before a meal
  Other Names: Glufast
  Arms: M
Drug: Voglibose — voglibose 0.2mg three times a day before a meal
  Other Names: Basen
  Arms: V

SUMMARY:
We will evaluate the efficacy and safety of combination therapy of 10 mg mitiglinide or 0.2mg voglibose with insulin glargine for 16 weeks after single administration of insulin glargine for 4 weeks in type 2 diabetic patients whose glycemic control were not enough despite administration of oral antidiabetic drug or insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* The type 2 diabetic patients aged between 30 and 70
* The patients whose Hb1Ac is over 7.0% despite administration of two or more oral antidiabetic drugs over 6 months or only insulin glargine over 3 months before registration
* Outpatients whose BMI is between 21 and 40 kg/㎡
* The patients who consented to participate in the clinical study in writing

Exclusion Criteria:

* The patients who have been using insulin formulation except insulin glargine
* The patients whose fasting blood glucose is over 270 mg/dL
* The patients whose C-peptide is under 1ng/ml on an empty stomach
* The patients who was surgically operated of gastrointestinal tract
* The patients who need additional treatment or who underwent operation within 3 months for severe complication such as diabetic foot ulcer, retinopathy and neuropathy
* The patients with severe hepatic dysfunction : uncompensated hepatic cirrhosis, or the case where aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is over 2.5 times higher than the normal limit ( ≥ 2.5 x normal ranges)
* The patients with unstable angina or acute myocardial infarction occurred within 3months
* The patients with renal failure or severe hypertension : diastolic blood pressure is over 110mmHg despite drug treatment
* The patients who have a life-threatening disease such as cancer or severe infection
* The patients with a history of drug allergy
* Pregnant or breast feeding or the women who are likely to be pregnant
* The patients who need oral or parenteral corticosteroids
* The patients who were judged to be unsuitable to the clinical study by other reasons

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c before and after administration of test drug | 20 weeks

SECONDARY OUTCOMES:
Change of self-monitoring of blood glucose before and after administration of test drug | 20 weeks
Change of insulin dose before and after administration of test drug | 20 weeks
Achievement rate of HbA1c target level (rate of the patients whose HbA1c were improved under 6.5% after administration) | 20 weeks
Change of CRP, 8-OHdG and Nitrotyrosine before and after administration of test drug | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kun-ho Yoon, Study Chair — The Catholic Univ. of Korea, Kangnam ST. Mary's Hospital
Locations (1):
- The Catholic Univ. of Korea, Kangnam ST. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Son JW, Lee IK, Woo JT, Baik SH, Jang HC, Lee KW, Cha BS, Sung YA, Park TS, Yoo SJ, Yoon KH. A prospective, randomized, multicenter trial comparing the efficacy and safety of the concurrent use of long-acting insulin with mitiglinide or voglibose in patients with type 2 diabetes. Endocr J. 2015;62(12):1049-57. doi: 10.1507/endocrj.EJ15-0325. Epub 2015 Sep 25. PMID 26411328